CLINICAL TRIAL: NCT05675111
Title: Endocrine-related Adverse Events Caused by Immune Checkpoint Inhibitors
Brief Title: Immune Checkpoint Inhibitors(ICPis)-Induced Endocrine Immune-related Adverse Events (irAEs)
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yang Tao, Chief, Department of Endocrinology & Metabolism The First Affiliated Hospital of Nanjing Medical University, Nanjing Medical University
Other Study IDs: 2020-SR-544.A1
Record Dates: First submitted 2023-01-01; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Immune Checkpoint Inhibitor; Endocrine Toxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Nanjing: The First Affiliated Hospital of Nanjing Medical University
- Zhengzhou: Henan Provincial People's Hospital
- Qingdao: The Affiliated Hospital of Qingdao University
- Urumqi: People' s Hospital of Xinjiang Uygur Autonomous Region
- Jinan: Shandong Provincial Hospital Affiliated to Shandong First Medical University

SUMMARY:
Immune checkpoint inhibitor (ICI) includes agents that block cytotoxic T-cell-associated antigen 4 (CTLA-4), programmed cell death protein 1 (PD-1), and programmed cell death protein ligand 1 (PD-L1). Since the FDA-approval of the CTLA-4 inhibitor ipilimumab in 2011, ICI drugs have emerged as a powerful new tool in the treatment for several advanced cancers. Now indications for ICI have expanded dramatically due to their efficacy and include a wide array of cancer types. However, the administration of ICI, whereas, carry the risk of developing immune-related adverse events (irAEs) and may lead to serious and even fatal events. Endocrine dysfunctions are among the most common irAEs that have been reported in clinical trials with ICI, including thyroid dysfunction, hypopituitarism, primary adrenal insufficiency (PAI) and insulin-deficient diabetes (ICI-DM). However, it is difficult to acquire a complete picture of irAEs from randomized controlled trials (RCTs) due to limitations in the study design and realistic practicalities.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients who received one dose or more of PD-1/PD-L1 inhibitors

Exclusion Criteria:

* Insufficient reported details
* Patients younger than 18 years old
* in a double-blind study where treatment allocation cannot be resolved

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older, with cancers who received one dose or more of PD-1/PD-L1 inhibitors 5 academic centers from June 2018 to March 2021 were included.
Sampling Method: Non-Probability Sample
Enrollment: 12408 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
irAEs | through study completion, an average of 2 year
  Immune Checkpoint Inhibitors Induced Endocrine Immune related Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Tao Yang, MD/PhD, Study Chair — First Affiliated Hospital, Nanjing Medical University
Locations (1):
- First Affiliated Hospital, Nanjing Medical University, Nanjing, Jiangsu, China